CLINICAL TRIAL: NCT05697991
Title: Non-Alcoholic Fatty Liver Disease in a Saudi Cohort With Type 2 Diabetes Mellitus
Acronym: CORDIAL
Status: Recruiting | Type: Observational
Sponsor: King Saud University (Other)
Collaborators: King Fahad Medical City (Other Government)
Responsible Party: Principal Investigator, Assim Alfadda, Prof., King Saud University
Other Study IDs: CORDIAL KSU
Record Dates: First submitted 2023-01-05; First posted 2023-01-26 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Nonalcoholic Fatty Liver Disease; Type 2 Diabetes Mellitus
Keywords: T2DM; Fatty Liver Disease; NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Biospecimen Retention: Samples With DNA — DNA, Serum, Urine and Stool

SUMMARY:
The global rise in the prevalence of obesity paved the way for the increased prevalence of yet another obesity-related complication significant enough to be considered within the roster of major public health threats: non-alcoholic fatty liver disease (NAFLD). In this follow-up study, the investigators will attempt to decipher the natural history of hepatic steatosis among patients with type 2 diabetes mellitus (T2DM) using state-of-the-art methods in a well-characterized Saudi cohort. The investigators aim also to validate existing biomarkers of disease severity and explore the pathogenesis of progressive disease using metabolic profiling technologies. A total of 1000 adult Saudi patients (males and females) with T2DM will be recruited. Those with co-morbidities, including hepatic decompensation, will be excluded. Participants will be followed three times for a total of 10 years/patient (Year 2, Year 5, and Year 10), and measures such as dietary evaluations, anthropometrics, and urine, stool, and blood examinations will be performed. Patients who develop NAFLD will be noted, and patterns/changes in the metabolic profile will be examined. For this specific grant (the first 2 years of the whole project), the investigators will be able to recruit the study cohort, do the baseline anthropometric, imaging, and biochemical measurements, and report the prevalence of NAFLD among patients with T2DM. This information will be the basis of subsequent follow-up and allow for validating potential diagnostic and prognostic biomarkers. This project will be of high importance at the national level since it will create awareness in the local medical community of the current severity status of NAFLD in the kingdom and will be used as a tool to promote public health awareness in the community.

DETAILED DESCRIPTION:
The increased prevalence of obesity in both the developed and developing worlds paved the way to the increased prevalence of yet another obesity-related complication significant enough to be considered within the roster of major public health threats: non-alcoholic fatty liver disease (NAFLD). It has been estimated that approximately 20% to 30% of the adult population harbors NAFLD. It is also the most common liver pathology among children of developed countries. Unfortunately, despite the alarming figures, NAFLD remains largely underdiagnosed, probably because of its less aggressive nature and benign presentation compared with other liver diseases. Thus, it is apparent that NAFLD, being a precursor to more serious liver conditions such as cirrhosis and hepatocellular carcinoma, should be given equal, if not greater, clinical significance.

Accumulating evidence has pointed to parallel clinical similarities between NAFLD and metabolic syndrome (MetS), the clustering of cardiovascular risk factors with insulin resistance as the common unifying factor. It is well established that persons with MetS are at greater risk of progressing to major chronic non-communicable diseases such as coronary artery disease and type 2 diabetes mellitus (T2DM). Consequently, patients with T2DM are more likely to develop NAFLD. Obesity is acknowledged as one of the common denominators linking NAFLD, MetS, and T2DM, making dietary and lifestyle modifications the gold standard for the treatment of these clinical entities aside from pharmacotherapy that aims to improve insulin sensitivity. Therefore, it is important to better understand the intricate pathophysiology of NAFLD among patients with T2DM so that future interventions will be aimed at reversing complications.

Our current knowledge of NAFLD in terms of prognosis and treatment is promising yet inconclusive, which means that further investigations using prospective approaches are required. Only recently was a consensus design for clinical trials and endpoints for non-alcoholic steatohepatitis (NASH) reported. In this follow-up study, the investigators attempt to decipher the natural history of hepatic steatosis among patients with T2DM using state-of-the-art methods in a well-characterized Saudi cohort. Diabetes, and its related medical complications, have been identified as one of the priority areas of the National Plan for Science and Technology in the Kingdom of Saudi Arabia (KSA).

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent prior to screening
* Men and women aged 18 to 60 years
* T2DM

Exclusion Criteria:

* Evidence of hepatic decompensation (ascites, clinical jaundice-bilirubin ≥ 40 µmol/L, encephalopathy)
* Preexisting hepatocellular carcinoma
* Other preexisting hepatic or extrahepatic malignancy
* Previous overt ischemic heart disease (myocardial infarction or acute coronary syndrome) or cerebrovascular disease (stroke or transient ischemic attack)
* Previous coronary artery bypass grafting, angioplasty, or stenting
* Any other issues that, in the opinion of the investigators, may preclude satisfactory completion of the study protocol

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population included patients who participated in the Cohort of Non-alcoholic Fatty Liver Disease with T2DM (the CORDIAL Study). This prospective cohort study started in 2015 and recruited patients from King Fahad Medical City (KFMC) and affiliated Primary Care Centers in Riyadh, Saudi Arabia. The patients will be prospectively followed up for 10 years for hepatic, metabolic, renal, and cardiovascular complications.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-03-23 (Actual); Primary Completion 2030-04-23 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of hepatic steatosis in T2DM | 15 years
  Fatty liver will be assessed by USS and FibroScan in patients with T2DM

SECONDARY OUTCOMES:
Progression of hepatic steatosis to advanced liver disease will be assessed by USS and FibroScan. | 15 years
  Assessment of hepatic steatosis progression to advanced liver disease by USS and FibroScan.
Pathogenesis of progressive disease | 15 years
  Untargeted metabolomics using a high-throughput proton NMR metabolomics approach for the screening of novel metabolites to understand the pathogenesis of progressive disease

CONTACTS AND LOCATIONS:
Overall Officials: Assim Alfadda, MD, Principal Investigator — King Saud University
Locations (1):
- King Fahad Medical City, Riyadh, Select A State Or Province, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
was not including in protocol and consent form

REFERENCES:
- [Derived] Alfadda AA, Alqutub AN, Sherbeeni SM, Aldosary AS, Alqahtani SA, Isnani A, Gul R, Khaleel MS, Alqasim SM, Almaghamsi AM. Predictors of liver fibrosis progression in cohort of type 2 diabetes mellitus patients with MASLD. J Diabetes Complications. 2025 Feb;39(2):108910. doi: 10.1016/j.jdiacomp.2024.108910. Epub 2024 Nov 20. PMID 39675110